CLINICAL TRIAL: NCT07312942
Title: Effects of Adding a Controlled Breathing Protocol to a Therapeutic Exercise Program in Adults With Multiple Myeloma
Brief Title: Effects of Controlled Breathing Added to Therapeutic Exercise in Multiple Myeloma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Isidro Fernández López, Principal Investigator, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Breathing Mieloma
Record Dates: First submitted 2025-12-17; First posted 2025-12-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma; Breathing Techniques; Breathing Exercises; Exercise Activity; Diaphragmatic Breathing
Keywords: Multiple myeloma; Breathing; Diaphragmatic breathing; Slow breathing; exercise activity; Breathing exercises
MeSH Terms: conditions — Multiple Myeloma; Respiratory Aspiration; Hypoventilation | interventions — Exercise Therapy

STUDY DESIGN:
Intervention Model Description: A randomized, parallel, double-blind, controlled, multicenter clinical trial with two intervention arms. Two groups of participants will be included, both receiving an educational session with a standardized educational leaflet on the importance of proper breathing, and a therapeutic exercise intervention over a 6-week period. One of the groups will additionally perform a home-based controlled breathing exercise protocol. Pre- and post-intervention assessments (6 weeks) will be conducted, along with a follow-up evaluation 4 weeks after completion of the intervention.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Only the principal investigator will have access to the randomization sequence, thereby maintaining blinding for the rest of the team involved in data collection.
  Both groups will receive the same therapeutic exercise program and an educational session with a standardized educational leaflet on the importance of physical activity and proper breathing in daily life, with the aim of minimizing differences in the perceived intervention.
  The study will include evaluator blinding, as all assessments will be carried out by an independent investigator who is not involved in the randomization process and is unaware of participants' group allocation. Additionally, statistical analyses will be conducted by a specialized statistician, also blinded to group assignment, thereby ensuring impartiality in the analysis and interpretation of the results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic exercise + initial educational session on proper breathing (Active Comparator): * Perform three weekly sessions of mobility and muscle-strengthening exercises (two on-site and one home-based) for 6 weeks. The home-based exercise program will consist of completing, once per week during the 6-week intervention, a structured session that replicates the logic and technique of the on-site program.
  * Walk a minimum of 7,000 steps/day or 50 minutes/day, three days per week.
  * To promote adherence to the protocol and standardize basic knowledge regarding the breathing technique, all participants will receive an initial educational session delivered on the first day of the on-site intervention. This session will include an introductory lecture and an explanatory leaflet outlining the fundamental principles of functional breathing and its relevance to the intervention.
  Interventions: Other: Therapeutic exercise + initial education session
- Therapeutic exercise + initial education session + home-based controlled breathing exercise protocol (Experimental): * Participants will perform a controlled breathing protocol at home twice daily, at least five days per week, throughout the 6-week study period, following the recommendations of the principal investigator.
  * Perform three weekly sessions of mobility and muscle-strengthening exercises (two on-site and one home-based) for 6 weeks. The home-based exercise program will consist of completing, once per week during the 6-week intervention, a structured session that replicates the logic and technique of the on-site program.
  * Walk a minimum of 7,000 steps/day or 50 minutes/day, three days per week.
  * To promote adherence to the protocol and standardize basic knowledge regarding the breathing technique, all participants will receive an initial educational session delivered on the first day of the on-site intervention. This session will include an introductory lecture and an explanatory leaflet outlining the fundamental principles of functional breathing and its relevance to the intervention.
  Interventions: Other: Controlled breathing exercise protocol + therapeutic exercise + initial education session

INTERVENTIONS:
Other: Controlled breathing exercise protocol + therapeutic exercise + initial education session — In addition to the therapeutic exercise protocol and the educational session on proper breathing, participants will perform a controlled breathing protocol at home twice daily, at least five days per week, throughout the 6-week study period, following the recommendations of the principal investigator. The goal is to integrate slow, gentle, diaphragmatic, nasal breathing into daily life.
  To promote adherence and ensure correct and consistent execution, participants will have access through the Web-App to two audio files containing guided breathing instructions and visualization exercises. These recordings were specifically developed for this project by a physiotherapist with more than 20 years of experience in respiratory control-based interventions, and were reviewed and approved by the entire research team.
  Other Names: Therapeutic exercise; educational session on proper breathing
  Arms: Therapeutic exercise + initial education session + home-based controlled breathing exercise protocol
Other: Therapeutic exercise + initial education session — In addition to the therapeutic exercise protocol and the educational session on proper breathing, participants will perform:
  -Three weekly sessions of mobility and muscle-strengthening exercises (two on-site and one home-based) for 6 weeks. The on-site sessions will last between 30 and 40 minutes and will take place at the Rehabilitation Department of Hospital 12 de Octubre in Madrid (a total of 12 on-site sessions-two per week). The home-based exercise program will consist of completing, once per week during the 6-week intervention, a structured session that replicates the logic and technique of the on-site program.
  A maximum of four absences from the on-site therapeutic exercise program will be allowed, and on those occasions the patient must register via the web application that they completed the prescribed home-based program.
  -Walk a minimum of 7,000 steps/day or 50 minutes/day, three days per week.
  Other Names: educational session on proper breathing; therapeutic exercise
  Arms: Therapeutic exercise + initial educational session on proper breathing

SUMMARY:
A randomized, parallel, double-blind, controlled, multicenter clinical trial with two intervention arms. Two groups of participants will be included, both receiving a therapeutic exercise intervention and an educational session on the importance of proper breathing over a 6-week period. One of the groups will additionally perform a home-based controlled breathing exercise protocol. Pre- and post-intervention assessments (6 weeks) will be conducted, along with a follow-up evaluation 4 weeks after completion of the intervention.

The goal is to determine the effectiveness of adding a controlled breathing exercise program to a therapeutic exercise intervention on somatic symptoms in individuals with multiple myeloma

DETAILED DESCRIPTION:
Randomized, parallel, double-blind, controlled clinical trial in which two groups of participants will be included and randomly assigned to one of the two intervention arms:

Therapeutic exercise + initial educational session on proper breathing.

Therapeutic exercise + initial educational session on proper breathing + home-based controlled breathing exercise protocol.

The therapeutic exercise and controlled breathing program will last 6 weeks. During this period, participants will:

Perform three weekly sessions of mobility and muscle-strengthening exercises (two on-site and one home-based) for 6 weeks. The on-site sessions will last between 30 and 40 minutes and will take place at the Rehabilitation Department of Hospital 12 de Octubre in Madrid (a total of 12 on-site sessions-two per week). The home-based exercise program will consist of completing, once per week during the 6-week intervention, a structured session that replicates the logic and technique of the on-site program.

Walk a minimum of 7,000 steps/day or 50 minutes/day, three days per week.

Perform a controlled breathing protocol twice per day at home during the 6-week study period, following the recommendations of the principal investigator. The goal is to integrate slow, gentle, diaphragmatic, nasal breathing into daily life.

The variables to be assessed will include: somatic symptom questionnaire, quality of life, sleep quality, fatigue, anxiety and depression symptoms.

These variables will be evaluated at baseline, at the end of the 6-week intervention period, and again 4 weeks after completing the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Confirmed diagnosis of multiple myeloma, currently undergoing active treatment with daratumumab, and under clinical follow-up by the Hematology Department of HU12O.
* Explicit medical indication for supervised physical activity issued by the responsible hematologist and documented in the medical record.
* No scheduled hematopoietic stem cell transplantation within the 60 days following the planned start date of the intervention (verified through medical record review).
* Functional status of ECOG 0-2 (Eastern Cooperative Oncology Group), assessed by a healthcare professional from the Hematology Department, ensuring the ability to perform at least basic and light instrumental activities of daily living, including independent ambulation.
* Access to a smartphone with stable internet connection, required for monitoring and recording adherence to the intervention.
* Ability to provide written informed consent, demonstrating understanding of the study's nature, purpose, and procedures.

Exclusion Criteria:

* Medical risk contraindicating exercise or breathing techniques:

  +Clinically significant cardiovascular disease, including: decompensated heart failure, acute myocardial infarction within the past 3 months, clinically uncontrolled arrhythmias, unstable angina, acute-phase deep vein thrombosis or pulmonary embolism, pacemakers or cardiac devices whose monitoring parameters contraindicate supervised exercise according to cardiology.
  * Severe decompensated respiratory disease, such as acute exacerbation of COPD, severe respiratory insufficiency, or persistently low resting oxygen saturation < 90% (not correctable).
* High musculoskeletal or bone risk:

  * Extensive lytic bone lesions, high risk of pathological fracture, or unstable vertebral fracture, documented by imaging or based on the assessment of the Hematology/Traumatology specialist.
  * Uncontrolled pain that prevents safe participation in an exercise program.
* Hematologic or systemic conditions contraindicating exercise:

  * Severe anemia: hemoglobin < 9 g/dL in women or < 8 g/dL in men (latest laboratory test ≤ 14 days).
  * Active systemic infection contraindicating exercise, fever ≥ 38 °C, or neutropenia < 0.5 × 10⁹/L.
  * Severe cytopenias that, in the opinion of the hematologist, preclude moderate exercise.
* Functional or procedural limitations:

  * Inability to remain in the supine position for ≥ 5 minutes, required for part of the breathing intervention.
  * Confirmed pregnancy or reasonable suspicion of pregnancy.
  * Severe cognitive impairment, major psychiatric disorders, or neurological diseases that limit understanding of the procedures or safe participation.
  * Significant difficulty understanding the language (spoken or written) that prevents following essential instructions or completing validated questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Somatic Symptom Questionnaire | Information for this variable will be collected at three time points: at baseline, at the end of the intervention (6 weeks), and four weeks after completion of the protocol.
  The PHQ-15 will be used to assess the number of somatic symptoms and the degree of distress experienced during the past four weeks. Cancer survivors with a greater number of somatic symptoms tend to report higher levels of stress, partly due to increased fear of disease recurrence or progressio

SECONDARY OUTCOMES:
Global quality of life | Information for this variable will be collected at three time points: at baseline, at the end of the intervention (6 weeks), and four weeks after completion of the protocol.
  Global quality of life will be assessed using the EORTC-QLQ C30 Version 3.0 questionnaire, developed by the European Organization for Research and Treatment of Cancer (EORTC), a cancer-specific instrument that has been extensively validated in both its English and Spanish versions
Sleep Quality Questionnaire | Information for this variable will be collected at three time points: at baseline, at the end of the intervention (6 weeks), and four weeks after completion of the protocol.
  The Pittsburgh Sleep Quality Index (PSQI) will be used in its validated Spanish version, which provides a global sleep quality score as well as partial scores across seven distinct components
Anxiety and Depression Scale | Information for this variable will be collected at three time points: at baseline, at the end of the intervention (6 weeks), and four weeks after completion of the protocol.
  The Hospital Anxiety and Depression Scale (HADS) will be used to assess these symptoms among study participants. This screening instrument has been widely used and validated as a brief tool for detecting depressive and anxiety symptoms in oncology patients

OTHER OUTCOMES:
Fatigue | Information for this variable will be collected at three time points: at baseline, at the end of the intervention (6 weeks), and four weeks after completion of the protocol.
  The Brief Fatigue Inventory (BFI) will be used to assess fatigue; it is a reliable instrument that allows for rapid evaluation of fatigue levels in cancer patients, and its Spanish version has also been validated

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Plaza-Manzano, PhD, Study Director — Department of Physiotherapy, Faculty of Nursing, Physiotherapy and Podiatry. Universidad Complutense de Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Shahriari M, Dehghan M, Pahlavanzadeh S, Hazini A. Effects of progressive muscle relaxation, guided imagery and deep diaphragmatic breathing on quality of life in elderly with breast or prostate cancer. J Educ Health Promot. 2017 Apr 19;6:1. doi: 10.4103/jehp.jehp_147_14. eCollection 2017. PMID 28546966
- [Background] Fournie C, Verkindt C, Dalleau G, Bouscaren N, Mohr C, Zunic P, Cabrera Q. Rehabilitation program combining physical exercise and heart rate variability biofeedback in hematologic patients: a feasibility study. Support Care Cancer. 2022 Mar;30(3):2009-2016. doi: 10.1007/s00520-021-06601-2. Epub 2021 Oct 12. PMID 34636946
- [Background] Dhruva A, Miaskowski C, Abrams D, Acree M, Cooper B, Goodman S, Hecht FM. Yoga breathing for cancer chemotherapy-associated symptoms and quality of life: results of a pilot randomized controlled trial. J Altern Complement Med. 2012 May;18(5):473-9. doi: 10.1089/acm.2011.0555. Epub 2012 Apr 23. PMID 22525009
- [Background] Shao R, Man ISC, Lee TMC. The Effect of Slow-Paced Breathing on Cardiovascular and Emotion Functions: A Meta-Analysis and Systematic Review. Mindfulness. 2024;15(1):1-18. doi:10.1007/s12671-023-02294-2
- [Background] Nicol JL, Chong JE, McQuilten ZK, Mollee P, Hill MM, Skinner TL. Safety, Feasibility, and Efficacy of Exercise Interventions for People With Multiple Myeloma: A Systematic Review. Clin Lymphoma Myeloma Leuk. 2023 Feb;23(2):86-96. doi: 10.1016/j.clml.2022.10.003. Epub 2022 Oct 22. PMID 36450625
- [Background] Moller MD, Ihorst G, Pahl A, Scheubeck S, Barsch F, Dold SM, Bertz H, Arends J, Wasch R, Engelhardt M. Physical activity is associated with less comorbidity, better treatment tolerance and improved response in patients with multiple myeloma undergoing stem cell transplantation. J Geriatr Oncol. 2021 May;12(4):521-530. doi: 10.1016/j.jgo.2020.11.003. Epub 2020 Nov 20. PMID 33223484
- [Background] Li J, Peng Y, Zhan D, Zhang Y, Yu S. Exercise interventions in patients with multiple myeloma: a scoping review. BMC Sports Sci Med Rehabil. 2025 Jun 9;17(1):148. doi: 10.1186/s13102-025-01193-4. PMID 40490782